CLINICAL TRIAL: NCT06473467
Title: Sedentaryism Triggered by Socio-economic Behavioral Changes During the Pandemic Period: the Overshadowed Danger
Brief Title: Socioeconomic Behavior Changes During the Pandemic
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Şensu Dinçer, MD, Istanbul University
Other Study IDs: sedentaryism
Record Dates: First submitted 2024-06-13; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Pandemic, COVID-19; Sedentary Behavior
Keywords: pandemic; socioeconomic behavioral changes; sedentaryism
MeSH Terms: conditions — COVID-19; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study was to determine the changing shopping and movement habits of people during the period of March 2020- June 2021, when full and partial lockdown measures were in force due to the covid 19 outbreak in our country. in 500 adult participants. The main questions were:

* whether the increase in sedentaryism that occurred during the pandemic will persist after the pandemic ended?
* whether the socioeconomic behavior patterns that emerged during the pandemic period will persist after the pandemic?

DETAILED DESCRIPTION:
A questionnaire was created by experts in order to examine the predicted changes with a numerical tool and on large audiences. Totally, 765 adult individuals (452 female, 313 male) answered the questionnaire. In the created questionnaire, it was envisaged to evaluate the changes by asking demographic data, shopping habits, exercise habits and health problems in the pre-closure period, closure period and post-closure period.

In order to determine the changing shopping habits of the participants, they were asked what type of shopping they did and how often, face to face and online, before the closure period (before March 2020), during the closure period (March 2020- June 2021) and after the closure period up to 2 years (June 2021-June 2023). A 5-point Likert scale was used to determine shopping frequency, with questions ranging from 1 for Never; and 5 for allways. Shopping types are listed as Daily Materials (Grocery Shopping), Clothing, Electronics, Cosmetics - Personal Care products, Household goods - Furniture, Ready-made food (Food ordering at home) and Gifts - Toys.

To determine the sedentary tendency of the participants, movement habits that distract from sedentary life were grouped under three headings. These were determined as weekly active sports activities, weekly non-sports activities that are expected to require movement, and the number of daily steps. In the prepared questionnaire, participants were asked before the closure period (before March 2020), during the closure period (March 2020- June 2021) and after the closure up to 2 years (June 2021-June 2023); which sports they engage in and their total active sports time; They were asked which non-sport activities they engaged in, their total non-sport activity time and daily step count.

In order to determine the health problems of the participants, if any, they were asked about the health problems they experienced before the closure period (before March 2020), during the closure period (March 2020- June 2021) and after the closure period up to 2 years (June 2021-June 2023).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* all genders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers aged 18 and over who agreed to participate in the study, were known by the authors from their workplace and home environment, and could be reached via email.
Sampling Method: Non-Probability Sample
Enrollment: 765 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
shopping habit (type) | before the closure period (before March 2020), during the closure period up to 2 years (March 2020- June 2021) and after the closure period (June 2021-June 2023)
  what type of shopping the participants did face to face and online.Shopping types are listed as Daily Materials (Grocery Shopping), Clothing, Electronics, Cosmetics - Personal Care products, Household goods - Furniture, Ready-made food (Food ordering at home) and Gifts - Toys.
shopping habit (frequency) | before the closure period (before March 2020), during the closure period (March 2020- June 2021) and after the closure period up to 2 years (June 2021-June 2023)
  A 5-point Likert scale was used to determine shopping frequency, with questions ranging from 1 for Never; and 5 for always.
sedantary score | before the closure period (before March 2020), during the closure period (March 2020- June 2021) and after the closure period up to 2 years (June 2021-June 2023)
  Participants were asked about their weekly active exercise times, weekly non-exercise activity times and daily step counts, and after the evaluation and scoring made in line with the answers given, it was determined which of the participants were closer to the sedentary lifestyle and which were farther away from the sedentary lifestyle.It was evaluated that participants with a total score of "5" and below were more prone to sedentary life, while participants with a score of "7" and above were more prone to active life.

CONTACTS AND LOCATIONS:
Locations (1):
- Şensu Dinçer, Istanbul, Turkey (Türkiye)